CLINICAL TRIAL: NCT04634123
Title: Evaluation Using of White Portland Cement and MTA in Pulpotomy Primary Anterior Teeth
Brief Title: The Use of Portland Cement in Primary Anterior Teeth Pulpotomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-Pedo-02-2021
Record Dates: First submitted 2020-01-31; First posted 2020-11-18 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Pulpotomies
Keywords: Pulpotomy; Portland cement; Primary Anterior Teeth

STUDY DESIGN:
Intervention Model Description: Split mouth design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary anterior teeth pulpotomy by White Portland Cement (Experimental)
  Interventions: Other: Pulpotomy therapy by White Portland Cement
- Primary anterior teeth pulpotomy by White MTA (Other)
  Interventions: Other: Pulpotomy therapy by White MTA

INTERVENTIONS:
Other: Pulpotomy therapy by White Portland Cement — Carious asymptomatic primary anterior teeth will be removed of dental caries likely to produce vital pulp exposure . The access will be refined using a sterile no. 4 or 6 round bur in a slow-speed handpiece . The remaining pulp will be treated using pulpotomy therapy by White Portland Cement
  Arms: Primary anterior teeth pulpotomy by White Portland Cement
Other: Pulpotomy therapy by White MTA — Carious asymptomatic primary anterior teeth will be removed of dental caries likely to produce vital pulp exposure . The access will be refined usinga sterile no. 4 or 6 round bur in a slow-speed handpiece . The remaining pulp will be treated using pulpotomy therapy by White MTA
  Arms: Primary anterior teeth pulpotomy by White MTA

SUMMARY:
- The aim of this study is to evaluate the effectiveness of White Portland cement and MTA in primary anterior teeth pulpotomy and follow up after 3 , 6 , 12 months ( Clinically and Radiographically) : Group A ( Control group ) : primary anterior teeth pulpotomized by White MTA . Group B : primary anterior teeth pulpotomized by White Portland Cement .

- The aim of this study is to evaluate the effectiveness of White Portland cement and MTA in pulpotomy primary canines for serial extraction and extract them after 3 months for Histopathlogic study : Group A ( Control group ) : primary canines pulpotomized by White MTA . Group B : primary canines pulpotomized by White Portland Cement .

DETAILED DESCRIPTION:
* Endodontic therapy for primary teeth faces several difficulties including morphology of root canals , physiological root absorption and failure to find ideal root-filling paste absorbs the same degree of root absorption .
* Pulpotomy therapy is considered easy , fast and does not include the length of canal or periapical region .
* The split mouth design will be adopted for the treated samples .
* Clinical success criteria :

  1. Absence of spontaneous or stimulant pain
  2. Absence gingival redness , swelling or fistula
  3. Physiological tooth mobility and absence sensitivity to percussion
* Radiographically success criteria :

  1. Absence periapical translucence
  2. Absence external or internal abnormal absorption

ELIGIBILITY:
Inclusion Criteria:

1. Age between 4 and 9 years.
2. Definitely positive or positive ratings of Frank scale.
3. Caries include maximum two surfaces
4. Pulp exposure during caries removal
5. Pulpal hemorrhage light red acceptable to hemostasis
6. Physiological root resorption no more than the apical third
7. Absence clinical and radiographic signs which indicate pulp necrosis

Exclusion Criteria:

1. Systematic or mental disorders.
2. Definitely negative or negative ratings of Frankel scale
3. Existence periapical translucence
4. Existence external or internal abnormal absorption
5. Existence swelling or fistula
6. Sensitivity to percussion
7. Existence of spontaneous or stimulant pain
8. Excessive movement

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of White Portland Cement pulpotomies 3 months after treatment | 3 months
  Clinical evaluation of White Portland Cement pulpotomies was performed 3 months after treatment using the preset clinical criteria. The pulpotomy procedure was decided a clinical success if the tooth fulfilled the following criteria: (1) No pain, (2) No swelling, (3) No tenderness to percussion, (4) No abscess or fistula, and (5) No abnormal tooth mobility
Clinical evaluation of White Portland Cement pulpotomies 6 months after treatment | 6 months
  Clinical evaluation of White Portland Cement pulpotomies was performed 6 months after treatment using the preset clinical criteria. The pulpotomy procedure was decided a clinical success if the tooth fulfilled the following criteria: (1) No pain, (2) No swelling, (3) No tenderness to percussion, (4) No abscess or fistula, and (5) No abnormal tooth mobility
Clinical evaluation of White Portland Cement pulpotomies 12 months after treatment | 12 months
  Clinical evaluation of White Portland Cement pulpotomies was performed 12 months after treatment using the preset clinical criteria. The pulpotomy procedure was decided a clinical success if the tooth fulfilled the following criteria: (1) No pain, (2) No swelling, (3) No tenderness to percussion, (4) No abscess or fistula, and (5) No abnormal tooth mobility
Clinical evaluation of White MTA pulpotomies 3 months after treatment | 3 months
  Clinical evaluation of White MTA pulpotomies was performed 3 months after treatment using the preset clinical criteria. The pulpotomy procedure was decided a clinical success if the tooth fulfilled the following criteria: (1) No pain, (2) No swelling, (3) No tenderness to percussion, (4) No abscess or fistula, and (5) No abnormal tooth mobility
Clinical evaluation of White MTA pulpotomies 6 months after treatment | 6 months
  Clinical evaluation of White MTA pulpotomies was performed 6 months after treatment using the preset clinical criteria. The pulpotomy procedure was decided a clinical success if the tooth fulfilled the following criteria: (1) No pain, (2) No swelling, (3) No tenderness to percussion, (4) No abscess or fistula, and (5) No abnormal tooth mobility
Clinical evaluation of White MTA pulpotomies 12 months after treatment | 12 months
  Clinical evaluation of White MTA pulpotomies was performed 12 months after treatment using the preset clinical criteria. The pulpotomy procedure was decided a clinical success if the tooth fulfilled the following criteria: (1) No pain, (2) No swelling, (3) No tenderness to percussion, (4) No abscess or fistula, and (5) No abnormal tooth mobility
Radiographic evaluation of White Portland Cement pulpotomies 3 months after treatment | 3 months
  Radiographic evaluation of White Portland Cement pulpotomies was performed 3 months after treatment using periapical radiographs. The pulpotomized tooth was judged to be radiographically successful if it demonstrated the following criteria: (1) Normal periodontal ligament space (2) No periapical and furcation pathosis, and (3) No internal resorption. If pulp canal obliteration (PCO) happened, it was recorded but not considered as a treatment failure
Radiographic evaluation of White Portland Cement pulpotomies 6 months after treatment | 6 months
  Radiographic evaluation of White Portland Cement pulpotomies was performed 6 months after treatment using periapical radiographs. The pulpotomized tooth was judged to be radiographically successful if it demonstrated the following criteria: (1) Normal periodontal ligament space (2) No periapical and furcation pathosis, and (3) No internal resorption. If pulp canal obliteration (PCO) happened, it was recorded but not considered as a treatment failure
Radiographic evaluation of White Portland Cement pulpotomies 12 months after treatment | 12 months
  Radiographic evaluation of White Portland Cement pulpotomies was performed 12 months after treatment using periapical radiographs. The pulpotomized tooth was judged to be radiographically successful if it demonstrated the following criteria: (1) Normal periodontal ligament space (2) No periapical and furcation pathosis, and (3) No internal resorption. If pulp canal obliteration (PCO) happened, it was recorded but not considered as a treatment failure
Radiographic evaluation of White MTA pulpotomies 3 months after treatment | 3 months
  Radiographic evaluation of White MTAt pulpotomies was performed 3 months after treatment using periapical radiographs. The pulpotomized tooth was judged to be radiographically successful if it demonstrated the following criteria: (1) Normal periodontal ligament space (2) No periapical and furcation pathosis, and (3) No internal resorption. If pulp canal obliteration (PCO) happened, it was recorded but not considered as a treatment failure
Radiographic evaluation of White MTA pulpotomies 6 months after treatment | 6 months
  Radiographic evaluation of White MTAt pulpotomies was performed 6 months after treatment using periapical radiographs. The pulpotomized tooth was judged to be radiographically successful if it demonstrated the following criteria: (1) Normal periodontal ligament space (2) No periapical and furcation pathosis, and (3) No internal resorption. If pulp canal obliteration (PCO) happened, it was recorded but not considered as a treatment failure
Radiographic evaluation of White MTA pulpotomies 12 months after treatment | 12 months
  Radiographic evaluation of White MTAt pulpotomies was performed 12 months after treatment using periapical radiographs. The pulpotomized tooth was judged to be radiographically successful if it demonstrated the following criteria: (1) Normal periodontal ligament space (2) No periapical and furcation pathosis, and (3) No internal resorption. If pulp canal obliteration (PCO) happened, it was recorded but not considered as a treatment failure
Histopathlogic evaluation of White Portland Cement 3 months after treatment | 3 months
  Histopathlogical evaluation of White Portland Cement pulpotomies was performed 3 months after treatment using the preset histopathlogical criteria. The pulpotomy procedure was decided a histopathlogical success if the tooth fulfilled the following criteria: (1) Normal soft tissue, (2) Formulation dentin bridge, (3) Normal bleeding from pulp tissue, (4) No fibrosis, and (5) No pulp calcification
Histopathlogic evaluation of White MTA 3 months after treatment | 3 months
  Histopathlogical evaluation of White MTA pulpotomies was performed 3 months after treatment using the preset histopathlogical criteria. The pulpotomy procedure was decided a histopathlogical success if the tooth fulfilled the following criteria: (1) Normal soft tissue, (2) Formulation dentin bridge, (3) Normal bleeding from pulp tissue, (4) No fibrosis, and (5) No pulp calcification

CONTACTS AND LOCATIONS:
Overall Officials: Hasan M Alzoubi, DDs, Principal Investigator — MSc student in Pedodontics, University of Damascus; Nada G Bshara, Phd, Study Director — Professor of Pedodontics, Department of Pedodontics, University of Damascus
Locations (1):
- Damascus Universite, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen TD, Judd PL, Barrett EJ, Sidhu N, Casas MJ. Comparison of Ferric Sulfate Combined Mineral Trioxide Aggregate Pulpotomy and Zinc Oxide Eugenol Pulpectomy of Primary Maxillary Incisors: An 18-month Randomized, Controlled Trial. Pediatr Dent. 2017 Jan 15;39(1):34-38. PMID 28292339
- [Background] Aminabadi NA, Farahani RM, Gajan EB. A clinical study of formocresol pulpotomy versus root canal therapy of vital primary incisors. J Clin Pediatr Dent. 2008 Spring;32(3):211-4. doi: 10.17796/jcpd.32.3.ghk26v4554790074. PMID 18524271
- [Background] Casas MJ, Kenny DJ, Johnston DH, Judd PL, Layug MA. Outcomes of vital primary incisor ferric sulfate pulpotomy and root canal therapy. J Can Dent Assoc. 2004 Jan;70(1):34-8. PMID 14709254
- [Background] Howley B, Seale NS, McWhorter AG, Kerins C, Boozer KB, Lindsey D. Pulpotomy versus pulpectomy for carious vital primary incisors: randomized controlled trial. Pediatr Dent. 2012 Sep-Oct;34(5):112-9. PMID 23211895
- [Background] Islam I, Chng HK, Yap AU. Comparison of the root-end sealing ability of MTA and Portland cement. Aust Endod J. 2005 Aug;31(2):59-62. doi: 10.1111/j.1747-4477.2005.tb00223.x. PMID 16128253